CLINICAL TRIAL: NCT00641771
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter 4-Week Study to Assess the Effect of Alendronate 70 mg and Vitamin D3 2800 IU Once Weekly on Fractional Calcium Absorption in Postmenopausal Osteoporotic Women
Brief Title: 4-Week Study to Assess the Effect of Alendronate and Vitamin D3 Once Weekly on Fractional Calcium Absorption in Postmenopausal Osteoporotic Women (0217A-230)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0217A-230; MK0217A-230; 2008_517
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MK0217A
  Interventions: Drug: alendronate sodium (+) cholecalciferol
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: alendronate sodium (+) cholecalciferol — MK0217A, a tablet containing alendronate 70-mg and vitamin D3 2800 IU, once weekly for 4 weeks. All patients will be instructed to take the tablet fasting upon arising for the day with 6 to 8 oz. of plain water (i.e., tap), wait at least one-half hour while continuing to fast and before the first food, beverage (except water), or other medication. All patients must eat before lying down.
  Other Names: MK0217A
  Arms: 1
Drug: Comparator: Placebo (unspecified) — MK0217A, Pbo tablet, once weekly for 4 weeks. All patients will be instructed to take the tablet fasting upon arising for the day with 6 to 8 oz. of plain water (i.e., tap), wait at least one-half hour while continuing to fast and before the first food, beverage (except water), or other medication. All patients must eat before lying down.
  Arms: 2

SUMMARY:
To compare change in fractional calcium absorption following administration of MK0217A relative to matching placebo, in postmenopausal women with osteoporosis

DETAILED DESCRIPTION:
Placebo will be administered over a 4 week, single-blind run-in phase. Calcium, as citrate-malate, will be administered throughout the study at an individualized dose supplementing the patient's daily dietary calcium intake to a total of approximately 1200 mg. At the end of the stabilization period, baseline calcium absorption will be determined and patients will be randomized to receive either MK0217A, or matching placebo once weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a postmenopausal osteoporotic female
* The patient is willing to limit direct sunlight exposure during the course of the study
* The patient must be ambulatory
* The patient has serum 25-hydroxyvitamin D =25 ng/mL

Exclusion Criteria:

* The patient is contraindicated to bisphosphonate therapy
* The patient has a vitamin D deficiency
* Patient will be excluded if their weight is above 85 kg
* The patient has a history of prior osteoporotic fracture
* The patient is currently or has received in the past treatment with effects on bone or calcium metabolism
* The patient has malabsorption syndrome
* The patient has active thyroid disease
* The patient has metabolic bone disease
* The patient had a myocardial infarction within 6 months of screening visit
* The patient has impaired renal function
* The patient is currently or has been a smoker in the last year

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-05; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To compare change in fractional calcium absorption following administration of MK0217A relative to matching placebo, in postmenopausal women with osteoporosis | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Shapses SA, Kendler DL, Robson R, Hansen KE, Sherrell RM, Field MP, Woolf E, Berd Y, Mantz AM, Santora AC 2nd. Effect of alendronate and vitamin D(3) on fractional calcium absorption in a double-blind, randomized, placebo-controlled trial in postmenopausal osteoporotic women. J Bone Miner Res. 2011 Aug;26(8):1836-44. doi: 10.1002/jbmr.395. PMID 21448918